CLINICAL TRIAL: NCT06959524
Title: AGENT DCB STANCE: AGENT Drug-Coated Balloon for STent AvoidANCE in PCI for De Novo Coronary Artery Disease
Brief Title: AGENT DCB STANCE: Safety and Effectiveness Study of AGENT Drug-Coated Balloon Compared to Standard of Care Percutaneous Coronary Intervention (PCI) Treatment for de Novo Coronary Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2530
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Arterial Disease (CAD); de Novo Lesions in Native Coronary Arteries
Keywords: Drug Coated Balloon; de novo; 97279374
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Masking Description: Where possible, independent outcome assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (8):
- Small Vessel - Test (Experimental): Small vessel subjects treated with AGENT DCB
  Interventions: Device: Drug Eluting Balloon
- Small Vessel - Control (Active Comparator): Small vessel subjects treated with drug eluting stent
  Interventions: Device: Drug eluting stent
- Bifurcation - Test (Experimental): Bifurcation subjects with side branches treated with AGENT DCB
  Interventions: Device: Drug Eluting Balloon
- Bifurcation - Control (Active Comparator): Bifurcation subjects with side branches treated with drug eluting stent or plain old balloon angioplasty
  Interventions: Device: Drug eluting stent; Procedure: Plain old balloon angioplasty
- Long Lesion - Test (Experimental): Long lesion subjects treated with AGENT DCB
  Interventions: Device: Drug Eluting Balloon
- Long Lesion - Control (Active Comparator): Long lesion subjects treated with drug eluting stent
  Interventions: Device: Drug eluting stent
- Overall - Test (Experimental): All subjects treated with AGENT DCB
  Interventions: Device: Drug Eluting Balloon
- Overall - Control (Active Comparator): All subjects treated with standard of care drug eluting stent and/or POBA
  Interventions: Device: Drug eluting stent; Procedure: Plain old balloon angioplasty

INTERVENTIONS:
Device: Drug Eluting Balloon — AGENT DCB
  Other Names: DCB
  Arms: Bifurcation - Test; Long Lesion - Test; Overall - Test; Small Vessel - Test
Device: Drug eluting stent — Any commercially available DES used for standard of care.
  Other Names: DES
  Arms: Bifurcation - Control; Long Lesion - Control; Overall - Control; Small Vessel - Control
Procedure: Plain old balloon angioplasty — Bifurcation side branch - POBA
  Arms: Bifurcation - Control; Overall - Control

SUMMARY:
AGENT DCB STANCE is a prospective, multicenter, open-label, 1:1 randomized controlled study designed to assess the safety and effectiveness of a treatment strategy with the AGENT Drug-Coated Balloon compared to standard of care percutaneous coronary intervention (PCI) treatment with drug eluting stent (DES) and/or balloon angioplasty in patients with de novo coronary lesions.

Subjects must have a de novo target lesion located in a native coronary artery.

DETAILED DESCRIPTION:
The study will also contain a PK sub study and an IVUS sub study.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed.
* Subject is eligible for percutaneous coronary intervention (PCI).
* Subject is willing to comply with all protocol-required follow-up evaluation.
* Women of child-bearing potential must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.

Angiographic Inclusion Criteria:

* Target lesion is a de novo lesion located in a native coronary artery
* Target lesion must have visually estimated stenosis > 50% and < 100% in symptomatic subjects (>70% and <100% in asymptomatic subjects) prior to lesion pre-dilation.
* Target lesion must be successfully pre-dilated.
* If a non-target lesion is treated, it must be treated first and must be deemed a success.

Clinical Exclusion Criteria:

* Subject has other serious medical illness (e.g. cancer, congestive heart failure) that may reduce life expectancy to less than 12 months.
* Subject has current problems with substance abuse (e.g. alcohol, cocaine, heroin, etc.).
* Subject has planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Subject is participating in another investigational drug or device clinical study that has not reached its primary endpoint.
* Subject intends to participate in another investigational drug or device clinical study within 12 months after the index procedure.
* Subject is a woman who is pregnant or nursing. A pregnancy test must be performed within 7 days prior to the index procedure, except for women who definitely do not have child-bearing potential.
* Subject has left ventricular ejection fraction known to be < 30%.
* Subject had PCI or other coronary interventions within the last 30 days.
* Subject has planned PCI or CABG after the index procedure.
* Subject had STEMI or QWMI <72h prior to the index procedure.
* Subject presents with NSTEMI and rising biomarkers, or ongoing chest pain or is hemodynamically unstable.
* Subject has cardiogenic shock (SBP < 80 mmHg requiring inotropes, IABP or fluid support).
* Subject has history (within 6 months prior to the index procedure) of New York Heart Association (NYHA) class III or IV heart failure.
* Subject is considered not able to tolerate at least 30 seconds of coronary occlusion of the target lesion.
* Subject has known allergy to paclitaxel or other components of the used medical devices.
* Subject has known hypersensitivity or contraindication to contrast dye that in the opinion of the investigator cannot be adequately pre-medicated.
* Subject has intolerance to antiplatelet drugs, anticoagulants required for procedure.
* Subject has platelet count < 100k/mm3 (risk of bleeding) or > 700k/mm3.
* Subject with renal insufficiency (creatinine ≥2.0 mg/dl) or failure (dialysis dependent).

Angiographic Exclusion Criteria:

* In-stent restenosis.
* Target lesion is located within a saphenous vein or arterial graft.
* Target lesion is a total occlusion or has evidence of thrombus present in the target vessel.
* Target lesion is severely calcified by angiography or has > 270° calcium arc on intravascular imaging or requires atherectomy.
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis) or three-vessel coronary disease requiring revascularization of all 3 vessels.
* Subject with planned treatment of lesion involving aortic ostial location.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1616 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate | 12-Month
  Target Lesion Failure (TLF) rate - defined as any ischemia-driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death. The MI events include the Peri-Procedural MI (PPMI) according to the SCAI MI definition and the spontaneous MI according to the 4th Universal MI definition.

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, Principal Investigator — Piedmont Heart Institute; Margaret McEntegart, Principal Investigator — NYPH/CUIMC
Locations (27):
- United States (25):
  - USC Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Pinnacle, Mechanicsburg, Pennsylvania
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
- Mater Private Hospital, Dublin, Ireland
- Clínico de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)